CLINICAL TRIAL: NCT06234020
Title: Frequency of Vertebro-spinal Anomalies in Patients Presenting With Ano-rectal Malformations
Brief Title: Frequency of Vertebrospinal Anomalies in Patients Presenting With Anorectal Malformations
Status: Completed | Type: Observational
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Mansoor Ahmed, Principal Investigator, Shaheed Zulfiqar Ali Bhutto Medical University
Other Study IDs: F.3-11/2023(ERRB)/Chairman
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Anorectal Malformations
MeSH Terms: conditions — Anorectal Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: To see the frequency of vertebrospinal anomalies in patients presenting with Anorectal Malformation — The patients presenting with anorectal malformation go through x-ray. We will get the reporting of x-ray done to see the vertebral anomalies and the patients presenting with fecal/urinary incontinence will go through MRI for spinal anomalies.

SUMMARY:
To determine the frequency of different vertebrospinal anomalies in patients with ARM

DETAILED DESCRIPTION:
106 pediatric patients presenting in Department of Neonatal and Paediatric Surgery, The Children Hospital, PIMS from date of approval up to 6 months with diagnosis of anorectal malforatioms will be enrolled in the study using non-probability convenience sampling technique. In this way, 106 patients will be included in the study. Patient selection will be made in the light of aforementioned exclusion and inclusion criteria of the study. Guardians of all patients will be explained about the study and informed consent will be obtained from them. Baseline data of enrolled patients will be recorded in the clinical questionnaire after careful history and examination. All patients born in our setup go through initial Xray of Lumbar spine and sacrum and ultrasound of spine which will be observed. Findings in the imaging will be noted in the clinical performa. It will be ensured that data is collected after approval of the synopsis and patient's confidentiality would not be breeched. Patients would have the autonomy to withdraw from study whenever they want.

ELIGIBILITY:
Inclusion Criteria:

* I.Neonates and Paediatric patients from age 1 day to 12 years II.Presenting in Department of Paediatric Surgery with Anorectal Malformation III.Both Pre and Post Op

Exclusion Criteria:

* Patients who have not consented for further investigations

Ages: 1 Day to 12 Years | Sex: All
Age Groups: Child
Study Population: Patients presenting in OPD, Emergency and admitted in ward.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
To determine the frequency of different vertebrospinal anomalies in patients with ARM | 6 months
  Following anomalies will be observed in patients of Anorectal Malformation:
  * Normal cord
  * Low lying conus
  * Thickened filum terminale
  * Tethered cord
  * Filum cyst
  * Vertebral anomalies
  * Borderline conus
  * Cervical rib (unilateral)
  * Cervical rib (bilateral)
  * Rudimentary 12th thoracic rib
  * Absent 12th thoracic rib
  * Lumbar rib
  * Syrinx
  * Ventriculus terminalis
  * Prominent central canal

CONTACTS AND LOCATIONS:
Locations (1):
- Shaheed Zulfiqar Ali Bhutto Medical University/PIMS, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No
Confidentiality